CLINICAL TRIAL: NCT03820063
Title: Image-guided De-escalation of Neo-adjuvant Chemotherapy in HER2-positive Breast Cancer: the TRAIN-3 Study
Acronym: TRAIN-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Borstkanker Onderzoek Groep (Network)
Collaborators: Roche Pharma AG (Industry); BOOG Study Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2018-01
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: neo adjuvant; HER2 positive; de-escalation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: neoadjuvant courses PTC-Ptz; adjuvant courses Ptz (pCR) or T-DM1 (non-pCR)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PTC-Pz (Experimental): * Paclitaxel 80mg/m2 administered intravenously on day 1 and day 8
  * Herceptin® 6mg/kg administered intravenously on day 1 (loading dose 8mg/kg) or Herceptin® administered subcutaneously 600mg on day 1
  * Carboplatin AUC 6mg•ml/min administered intravenously on day 1
  * Pertuzumab 420mg administered intravenously on day 1 (loading dose 840mg)
  * Treatment cycles are repeated on day 22
  Patients who do not achieve pCR will complete a total of nine cycles taxane-containing chemotherapy followed by 14 cycles of treatment with adjuvant T-DM1.
  Interventions: Drug: PTC-Pz

INTERVENTIONS:
Drug: PTC-Pz — * Paclitaxel 80mg/m2 administered intravenously on day 1 and day 8
  * Herceptin® 6mg/kg administered intravenously on day 1 (loading dose 8mg/kg) or Herceptin® administered subcutaneously 600mg on day 1
  * Carboplatin AUC 6mg•ml/min administered intravenously on day 1
  * Pertuzumab 420mg administered intravenously on day 1 (loading dose 840mg)
  * Treatment cycles are repeated on day 22
  In case of non pCR; Adjuvant T-DM1, 3.6mg/kg Q 22 days, for 14 cycles.

SUMMARY:
This is a multicenter, single arm, phase II study evaluating the efficacy of image-guided de-escalating neoadjuvant treatment with paclitaxel, Herceptin® (trastuzumab), carboplatin, and pertuzumab (PTC-Ptz) in stage II-Ill HER2-positive breast cancer.

DETAILED DESCRIPTION:
High pathological complete response (pCR)-rates are seen using different neoadjuvant chemotherapy schedules with trastuzumab and pertuzumab in HER2-positive stage II - III breast cancer patients. Total pCR rates in breast and axilla have been described as high as 64%, and with an even higher rate of >80% in patients with HER2-positive and hormone receptor (HR) negative tumors. PCR is associated with better long-term outcomes in patients with HER2-positive breast cancer. Three year progression-free survival ranges between 85-90%. Neoadjuvant treatment of HER2-positive breast cancer typically consists of six to nine cycles of treatment. Longer duration of treatment is associated with higher pCR-rates but gives more toxicity. Pathological complete responses are sometimes seen after only 10-12 days of neoadjuvant treatment. It is therefore important to investigate which patients can safely be treated with less than six cycles of chemotherapy and who requires more than six cycles for maximum activity.

The radiologic response of a breast tumor after neoadjuvant therapy is predictive of the pathologic response, although the accuracy differs between breast cancer subtypes. It is hypothesized that patients with an early complete radiologic response may not benefit from additional chemotherapy and can be referred for early surgery. Patients who have not achieved pCR after early surgery despite radiologic complete response (rCR) are candidates for further adjuvant chemotherapy to complete the initially planned number of treatment cycles and maintain maximum treatment activity. Imaged guided de-escalation in which the number of treatment cycles is determined by the radiologic response could thus reduce toxicity in neoadjuvant treatment while maintaining activity.

This study will evaluate the efficacy of image-guided de-escalation of neoadjuvant chemotherapy in patients with HER2-positive breast cancer.

To maintain efficacy, patients who do not achieve pCR will complete a total of nine cycles taxane-containing chemotherapy followed by 14 cycles of treatment with adjuvant T-DM1. Patients who achieve early pCR will continue treatment with Herceptin® and pertuzumab to complete one full year of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primairy infiltrating breast cancer.
2. Stage II or Ill disease.
3. Overexpression and/or amplification of HER2 in an invasive component of the core biopsy.
4. Age <:18
5. ECOG Group performance status
6. LVEF >50% measured by echocardiography, MRI or MUGA
7. Known HR-status ( in percentages)

Exclusion Criteria:

1. Previous radiation therapy of chemotherapy
2. Pregnancy or breastfeeding
3. Evidence of distant metastases
4. Evidence of bilateral infiltrating breast cancer
5. Concurrent anti-cancer treatment or another investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival at three years | 3 years
  Number of patients without progression of disease recurrence, second primary or death

SECONDARY OUTCOMES:
Overall survival at three years | 3 years
  Number of patients alive at three years
Pathologic complete response in breast and axilla | an average of 6 months
  Number of patients with absence of invasive tumor cells in breast and axilla at surgery
Radiologic complete response | an average of 6 months
  Number of patients with absence of pathologic enhancement on MRI
Number of neoadjuvant chemotherapy cycles administered | an average of 1 year
  Number of neoadjuvant chemotherapy cycles administered per patient
Number of radical and non-radical resections | an average of 6 months
  Number of patients with radical and non-radical resections
Incidence and severity of adverse events | an average of 1 year
  Number of patients with toxicity grade >= 3 (CTCAE v5.0) until 30 days after last adjuvant administration
Incidence and severity of cardiotoxicity and neuropathy | an average of 1 year
  Number of patients with cardiotoxicity and neuropathy grade >= 2 (CTCAE v5.0) until 30 days after last adjuvant administration
Incidence of symptomatic LVSD (heart failure), | an average of 1 year
  Number of patients with an asymptomatic decline in LVEF requiring treatment or leading to discontinuation of pertuzumab and Herceptin, or a decrease ≥10 percentage points from baseline to a LVEF <50%
Grade ≥3 laboratory test abnormalities | an average of 1 year
  Number of patients with Grade ≥3 laboratory test abnormalities
Incidence of number of tumor positive Vacuum Assisted Core Biopsy | an average 6 months
  Number of patients with tumor present at Vacuum Assisted Core Biopsy at the moment of radiological complete response on MRI

CONTACTS AND LOCATIONS:
Overall Officials: G S Sonke, MD, Principal Investigator — NKI-AvL; A E van Leeuwen- Stok, PhD, Study Director — BOOG Study Center
Locations (52):
- Netherlands (52):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - Amsterdam UMC, Amsterdam
  - NKI-AVL, Amsterdam
  - OLVG, Amsterdam
  - Gelre ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - Alexander Monro ziekenhuis, Bilthoven
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Groep, Delft
  - Deventer ziekenhuis, Deventer
  - van Weel Bethesda, Dirksland
  - Nij Smellinghe, Drachten
  - Ziekenhuisvoorziening Gelderse Vallei, Ede
  - Catharina ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Sint Annaziekenhuis, Geldrop
  - RIVAS Beatrixziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - Martini ziekenhuis, Groningen
  - Ziekenhuis St. Jansdal, Harderwijk
  - Tjongerschans, Heerenveen
  - Zuyderland Medisch Centrum, Heerlen
  - Elkerliek ziekenhuis, Helmond
  - Tergooi, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - MUMC, Maastricht
  - Sint Antonius ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Bernhoven, Oss
  - Stichting ziekenhuizen West-Friesland en Waterland, Purmerend
  - Laurentius ziekenhuis, Roermond
  - Erasmus MC, Universitair Medisch Centrum Rotterdam, Rotterdam
  - Franciscus Gasthuis en Vlietland, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Maasstadziekenhuis, Rotterdam
  - ZorgSaam, Terneuzen
  - Haaglanden MC, The Hague
  - Haga Ziekenhuis, The Hague
  - Rivierenland Ziekenhuis, Tiel
  - Elisabeth TweeSteden ziekenhuis, Tilburg
  - Diakonessenhuis Utrecht, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCurie Medisch Centrum voor Noord-Limburg, Venlo
  - SKB Ziekenhuis Winterswijk, Winterswijk
  - Zaans Medisch Centrum, Zaandam
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] van der Voort A, Louis FM, van Ramshorst MS, Kessels R, Mandjes IA, Kemper I, Agterof MJ, van der Steeg WA, Heijns JB, van Bekkum ML, Siemerink EJ, Kuijer PM, Scholten A, Wesseling J, Vrancken Peeters MTFD, Mann RM, Sonke GS; Dutch Breast Cancer Research Group. MRI-guided optimisation of neoadjuvant chemotherapy duration in stage II-III HER2-positive breast cancer (TRAIN-3): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2024 May;25(5):603-613. doi: 10.1016/S1470-2045(24)00104-9. Epub 2024 Apr 5. PMID 38588682